CLINICAL TRIAL: NCT00880243
Title: Effect of Priming With Granulocyte-Macrophage Colony-Stimulating Factor During Chemotherapy and Comparison of Timed Sequential Chemotherapy vs 4 Courses of High Dose Cytarabine as Consolidation in Younger Adults With Newly Diagnosed AML
Brief Title: Effect of Priming During Induction and Consolidations in Younger Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Acute Leukemia French Association (Other)
Collaborators: Hospices Civils de Lyon (Other)
Responsible Party: Xavier THOMAS, MD, PhD, Service Hematologie, LYON, France
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALFA 9802
Record Dates: First submitted 2009-04-08; First posted 2009-04-13 (Estimated); Last update posted 2009-04-13 (Estimated); Status verified 2009-04

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute myeloid leukemia; Priming; GM-CSF; Timed-sequential chemotherapy; Prognosis
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Granulocyte-Macrophage Colony-Stimulating Factor; Mitoxantrone; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- EMA+GM-CSF (Experimental): * Daunorubicine (CérubidineR) : 80 mg/m2/jour IV over 30 min from day 1 to day 3,
  * AraC (AracytineR) : 500 mg/m2/jour IV from day 1 to day 3,
  * Mitoxantrone (NovantroneR) : 12 mg/m2/jour IV over 30 min from day 8 to 9
  * AraC (AracytineR) : 500 mg/m2/12h IV over 3 hours from day 8 to day10.
  * GM-CSF (LeucomaxR): 5 µg/kg/jour IV over 6 hours from day 1 to day 10.
  Interventions: Drug: GM-CSF
- EMA without GM-CSF (Active Comparator): * Daunorubicine (CérubidineR) : 80 mg/m2/jour IV over 30 min from day 1 to day 3,
  * AraC (AracytineR) : 500 mg/m2/jour IV from day 1 to day 3,
  * Mitoxantrone (NovantroneR) : 12 mg/m2/jour IV over 30 min from day 8 to 9
  * AraC (AracytineR) : 500 mg/m2/12h IV over 3 hours from day 8 to day10.
  Interventions: Drug: GM-CSF
- HD AraC+ GM-CSF (Experimental): * AraC (Aracytine) : 3 g/m2/12h IV (3 hours) on days 1, 3 , 5
  * GM-CSF :5 µg/kg/d IV (6 hours) from day1 to day 5
  Interventions: Drug: GM-CSF
- HD-AraC without GM-CSF (Active Comparator): - AraC (Aracytine) : 3 g/m2/12h IV (3 hours) on days 1, 3 , 5
  Interventions: Drug: GM-CSF

INTERVENTIONS:
Drug: GM-CSF — Randomization 1: GM-CSF (5micogram/Kg/d) versus no GM-CSF during induction chemotherapy and all consolidation courses.
  Randomiization 2: Consolidation high dose AraC versus consolidation EMA
  Other Names: GM-CSF: molgramostim; AraC: Cytarabine; Daunorubicine: Cerubidine; EMA: etoposide, mitoxantrone, cytarabine

SUMMARY:
The purpose of this study is:

1. To compare priming with Granulocyte-Macrophage Colony-Stimulating Factor (GM-CSF) during induction and consolidation courses versus no priming.
2. To compare as consolidation timed sequential chemotherapy versus four courses of high dose cytarabine.

DETAILED DESCRIPTION:
Patients aged 15-50 are enrolled and randomly assigned to receive GM-CSF or no GM-CSF during all remission-induction and consolidation courses of chemotherapy. Induction chemotherapy consists of a timed-sequential chemotherapy including a first sequence of chemotherapy combining daunorubicin, 80 mg/m2 per day, administered IV as a short infusion over 3 days (days 1-3), and cytarabine, 500 mg/m2 per day IV as a continuous infusion over the same period. The second sequence, administered after 4-day free interval, consists of mitoxantrone, 12 mg/m2 per day, administered IV as a short infusion over 2 days (days 8 and 9), and cytarabine, 500 mg/m2/12h, administered as a 3-hour infusion for 3 days (days 8-10). Salvage therapy consists of cytarabine, 3 g/m2/12h on days 1,3,5,7, combined with amsacrine, 100mg/m2 per day on days 1 to 3. GM-CSF (Leucomax, recombinant human GM-CSF from Escherichia Coli, Schering Plough, Kenilworth,N.J., USA) is given at a dose of 5µg/kg per day, intravenously beginning at day 1 of each chemotherapy course and continuing until the last day of chemotherapy of each course.

Patients who achieve CR after induction chemotherapy or salvage therapy are randomly assigned to consolidation courses consisting of either a timed sequential chemotherapy similar to that of the ALFA-9000 trial (P2 arm) or the CALGB postremission chemotherapy (P1 arm), which includes 4 cycles of high-dose cytarabine, followed by 4 additional maintenance courses.

ELIGIBILITY:
Inclusion Criteria:

* A morphologically proven diagnosis of AML according to the WHO classification
* Serum creatinine < 2N; AST and ALT < 2.5N; total bilirubin < 2N (unless related to the underlying disease).
* ECOG performance status 0 to 2.
* Women of child-bearing must use acceptable contraceptive methods, and must have a negative serum or urine pregnancy test within 2 weeks prior the beginning treatment on this trial.
* Must be able and willing to give written informed consent

Exclusion Criteria:

* Patients with M3-AML. Patient with AML following diagnosed myeloproliferation or patient with prior history of MDS known for more than 3 months. Patients with AML secondary to previous treatment with cytotoxic chemotherapy or radiotherapy (therapy-related AML).
* Patient presenting any diagnosis of uncontrolled or metastatic tumor.
* Patients with uncontrolled severe infection,

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 473 (Actual)
Dates: Start 1999-03; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Assessing the potential value of the daily administration of GM-CSF during induction chemotherapy and post-induction for analyzing and comparing the arms with and without GM-CSF: EFS, % of CR, duration of remission, OS and toxicity of each treatment. | 72 months

SECONDARY OUTCOMES:
Evaluate the effectiveness on DFS of a single course of consolidation using a very intensive sequential chemotherapy with mitoxantrone, AraC and etoposide feasible compared to 4 courses of high dose AraC followed of 4 courses of maintenance. | 72 months

CONTACTS AND LOCATIONS:
Overall Officials: XAVIER THOMAS, MD, PhD, Principal Investigator — Hospices Civils de Lyon

REFERENCES:
- [Result] Thomas X, Raffoux E, Botton Sd, Pautas C, Arnaud P, de Revel T, Reman O, Terre C, Corront B, Gardin C, Le QH, Quesnel B, Cordonnier C, Bourhis JH, Elhamri M, Fenaux P, Preudhomme C, Michallet M, Castaigne S, Dombret H. Effect of priming with granulocyte-macrophage colony-stimulating factor in younger adults with newly diagnosed acute myeloid leukemia: a trial by the Acute Leukemia French Association (ALFA) Group. Leukemia. 2007 Mar;21(3):453-61. doi: 10.1038/sj.leu.2404521. Epub 2007 Jan 25. PMID 17252021
- [Derived] Thomas X, Elhamri M, Raffoux E, Renneville A, Pautas C, de Botton S, de Revel T, Reman O, Terre C, Gardin C, Chelghoum Y, Boissel N, Quesnel B, Hicheri Y, Bourhis JH, Fenaux P, Preudhomme C, Michallet M, Castaigne S, Dombret H. Comparison of high-dose cytarabine and timed-sequential chemotherapy as consolidation for younger adults with AML in first remission: the ALFA-9802 study. Blood. 2011 Aug 18;118(7):1754-62. doi: 10.1182/blood-2011-04-349258. Epub 2011 Jun 20. PMID 21690555
- [Derived] Boissel N, Nibourel O, Renneville A, Gardin C, Reman O, Contentin N, Bordessoule D, Pautas C, de Revel T, Quesnel B, Huchette P, Philippe N, Geffroy S, Terre C, Thomas X, Castaigne S, Dombret H, Preudhomme C. Prognostic impact of isocitrate dehydrogenase enzyme isoforms 1 and 2 mutations in acute myeloid leukemia: a study by the Acute Leukemia French Association group. J Clin Oncol. 2010 Aug 10;28(23):3717-23. doi: 10.1200/JCO.2010.28.2285. Epub 2010 Jul 12. PMID 20625116